CLINICAL TRIAL: NCT04146142
Title: A Prospective Randomized Trial of Antibiotic Prophylaxis Versus None Before Transperineal MRI-TRUS Fusion Guided Prostate Biopsy
Brief Title: Transperineal MRI-TRUS Fusion Guided Prostate Biopsy With vs Without Antibiotic Prophylaxis
Acronym: NORAPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Eduard Baco, Principal investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019/1266
Record Dates: First submitted 2019-10-28; First posted 2019-10-31 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Prostate Biopsy; Antibiotic
Keywords: Prostate Cancer; Biopsy; Complication; Randomization
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Antibiotic Prophylaxis

STUDY DESIGN:
Intervention Model Description: Randomized study 1:1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transperineal prostate biopsy with antibiotic profylaxis (Active Comparator): Cefuroxim 1.5 g will be applied intramuscularly before prostate biopsy
  Interventions: Procedure: Transperineal prostate biopsy with or without antibiotic prophylaxis
- Transperineal prostate biopsy without antibiotic profylaxis (Experimental): No antibiotics will be used before or after prostate biopsy
  Interventions: Procedure: Transperineal prostate biopsy with or without antibiotic prophylaxis

INTERVENTIONS:
Procedure: Transperineal prostate biopsy with or without antibiotic prophylaxis — As described above.

SUMMARY:
Prostate biopsy is indicated in patients with suspected prostate cancer and has been traditionally performed through the rectum using antibiotic prophylaxis. Increasing antibiotic resistance of intestinal bacteria is causing a growing number of patients to get post-biopsy infections. Sepsis rate after transrectal biopsies is approximately 4-10%.

To reduce the risk of post-biopsy infections, transperineal approach in general anesthesia and antibiotic prophylaxis has been used. The investigators at Oslo University Hospital Aker developed MRI -TURS elastic image fusion guided transperineal prostate biopsy technique in local anesthesia and Bactrim prophylaxis as outpatient procedure. The investigators found 0.4% post-biopsy infection rate. Afterwards a pilot study using the same biopsy technique however without antibiotic prophylaxis was realized in 90 patients. None of these subjects experienced infection.

The investigators wish to perform a prospective randomized trial of antibiotic prophylaxis versus none before transperineal MRI-TRUS fusion guided prostate biopsy in local anesthesia in outpatient clinic.

DETAILED DESCRIPTION:
Background: Unnecessary use of antibiotics promotes antibiotic resistance. Efforts for antibiotic use reduction without increase the risk of serious infection complications are therefore needed.

Purpose: The aim of this trial is to compare the rates of infectious complication after transperineal prostate biopsy in patients with and without antibiotic prophylaxis.

Materials and methods: A total of 450 patients will be included in this trial. A 1:1 randomization to receive or not receive antibiotics prophylaxis will be performed using randomization system WebCRF-3 system. MRI-TRUS fusion prostate biopsy will be done with transperineal prostate approach in local anesthesia in outpatient clinic. In patients with normal MRI,12-core systematic prostate biopsies with 3D biopsy registration will be done according to the EAU guidelines. In patients with positive MRI, 2-4 targeted biopsies from the suspicious MRI areas will be realized and systematic prostate biopsies will also be done. All prostate biopsies will be performed using Koelis MRI-TRUS image fusion and organ based tracking system. Post-biopsy infection and any adverse events will be systematically prospectively registered in all patients. Pain during the local anesthesia application and during the biopsy procedure will be registered using Visual Analog Score, 10 points scale questionnaire.

ELIGIBILITY:
Inclusion Criteria: Clinical indication for prostate cancer

-

Exclusion Criteria:

* Patients with symptoms of urinary tract infection or positive findings on urine dipstic before biopsy
* Patients with indwelling urethral catheter
* Patients with immunodeficiency disorders
* Patients with high risk for infective endocarditis [European Society of Cardiology]

  1. Patients with a prosthetic aortic or pulmonary valve
  2. Patients with previous infective endocarditis
  3. Patients with congenital heart disease who are cyanotic and those who have had palliative shunts/conduits/other prostheses
* Patients with a history of thromboembolic disease
* Patients with a history of allergy to the study drug
* Patients who do not wish to participate in the study

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 550 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence of sepsis | Up to 30 days
  Post biopsy sepsis will be defined by SIRS criteria
Incidence of post biopsy urinary tract infection | Up to 30 days
  Post biopsy urinary tract infection not demanding hospital admission within 30

OTHER OUTCOMES:
Pain during the local anesthesia application | Immediately after the intervention
  Patients will be asked to mention the intensity of pain during the anesthesia using Visual Analog Score for pain, range: 0 to 10, the worse is 10.
Pain during the prostate biopsy | Immediately after the intervention
  Patients will be asked to mention the intensity of pain during the prostate biopsy using Visual Analog Score for pain, range: 0 to 10, the worse is 10.

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Baco, MD, PhD, Principal Investigator — Oslo University Hospital, Oslo, Norway; Erik Rud, MD,PhD, Study Chair — Oslo University Hospital, Oslo, Norway; Karsten Gunzel, MD, Study Chair — Vivantes Klinkum Am Urban, Berlin, Germany
Locations (2):
- Vivantes Klinikum am Urban, Berlin, Germany
- Oslo University Hospital, Aker, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
All data generated during this study will be evaluated at Oslo University Hospital

REFERENCES:
- [Derived] Jacewicz M, Rud E, Lauritzen P, Baco E. Non-infectious adverse events of transperineal prostate biopsies performed under local anaesthesia. BJU Int. 2024 Aug;134(2):300-306. doi: 10.1111/bju.16383. Epub 2024 Apr 28. PMID 38679416
- [Derived] Jacewicz M, Gunzel K, Rud E, Sandbaek G, Magheli A, Busch J, Hinz S, Baco E. Antibiotic prophylaxis versus no antibiotic prophylaxis in transperineal prostate biopsies (NORAPP): a randomised, open-label, non-inferiority trial. Lancet Infect Dis. 2022 Oct;22(10):1465-1471. doi: 10.1016/S1473-3099(22)00373-5. Epub 2022 Jul 12. PMID 35839791